CLINICAL TRIAL: NCT02644993
Title: Registry for Analysis of Quality of Life, Normal Organ Toxicity and Survival of Pediatric Patients Treated With Proton Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Do Hoon Lim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-10-111
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Pediatric Cancer Patients
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton beam therapy (Experimental)
  Interventions: Radiation: Proton therapy

INTERVENTIONS:
Radiation: Proton therapy

SUMMARY:
The study aim of this study is to evaluate the effect of proton therapy on quality of life and long-term normal tissue toxicities of the pediatric cancer patients. Based on these results, the predictive model of long-term normal tissue toxicities, survival, and quality of life could be recognized. Risk-adapted treatment strategy based on the predictive model in pediatric cancer patients could be established.

ELIGIBILITY:
Inclusion Criteria:

* less than 18 years of age
* patient who is planned to receive proton therapy at Samsung Medical Center
* Informed consent

Exclusion Criteria:

* Refuse to participate this cohort study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | within 2 weeks before proton beam therapy

SECONDARY OUTCOMES:
Quality of Life Questionnaire baseline | within 1 week before proton beam therapy completion
Quality of Life Questionnaire | 3-6 months after proton beam therapy
Quality of Life Questionnaire | 1 year after proton beam therapy
Quality of Life Questionnaire | 3 years after proton beam therapy
Quality of Life Questionnaire | 5 years after proton beam therapy
Quality of Life Questionnaire | 10 years after proton beam therapy
Adverse event | 3-6 months after proton beam therapy
Adverse event | 1 year after proton beam therapy
Adverse event | 3 years after proton beam therapy
Adverse event | 5 years after proton beam therapy
Adverse event | 10 years after proton beam therapy

CONTACTS AND LOCATIONS:
Overall Officials: Do Hoon Lim, MD, PhD, Principal Investigator — Proton therapy center, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea